CLINICAL TRIAL: NCT00544531
Title: The Cytogenetic Constitution of Embryos Resulting From Immature Oocytes (M1)
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 76/05
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2005-09

CONDITIONS: Infertility
Keywords: MI oocytes, FISH,chromosomal aberrations
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the chromosomal number content in the blastomeres of embryos achieved from fertilization of immature oocytes at MI stage recruited following COH for IVF.

comparison of the genetic number content of embryos and their quality in terms of cleavage rate and morphological score reached after fertilization of immature oocytes at MI stage whether arrested at the MI stage or extruded the polar body, after in vitro maturation for a variable length of time.

DETAILED DESCRIPTION:
Patients undergoing routine IVF, following informed consent, donated some of their unusable, immature- MI stage oocytes for our research. Following in vitro maturation for up to 2, 4, 8 and 24 hours after harvest, all immature oocytes in these 4 study groups underwent intracytoplasmic donor sperm injection (ICSI), whether they extruded their polar body (MI-PB or rescued MI) or not (arrested MI). Oocyte fertilization rate after 24 hours and embryonic development in terms of cleavage rate and morphology were assessed, for another 48 hours. Then the whole embryo was prepared for molecular cytogenetic evaluation using FISH (Fluorescence in situ hybridization) analysis of chromosomes x, y and 18.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presence of immature oocytes after ART stimulation

Exclusion Criteria:

* Patients with less than total 7 oocytes

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23907 (Actual)
Dates: Start 2005-10; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ron-el, professor, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Infertility unit,Assaf-Harofeh Medical Center, Zrifin, Israel